CLINICAL TRIAL: NCT06350123
Title: A Phase IIb, Multicenter, Randomised, Double-Blind, Dose-finding Study to Evaluate the Efficacy, Safety and Tolerability of Balcinrenone in Combination With Dapagliflozin Compared With Dapagliflozin in Patients With Chronic Kidney Disease and Albuminuria
Brief Title: Efficacy, Safety and Tolerability of Balcinrenone/Dapagliflozin Compared to Dapagliflozin in Adults With Chronic Kidney Disease
Acronym: MIRO-CKD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6405C00002; 2023-509709-63-00 (Registry Identifier: EU CT number)
Record Dates: First submitted 2024-04-02; First posted 2024-04-05 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Multicentre, randomised, double-blind, dose-finding, parallel group, double-dummy
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Balcinrenone/dapagliflozin 15 mg/10 mg (Experimental): Patients will be randomized 1:1:1 to either balcinrenone/dapagliflozin and matching placebo for dapagliflozin or dapagliflozin and matching placebo for balcinrenone/dapagliflozin
  Interventions: Drug: Balcinrenone/dapagliflozin 15 mg/10 mg and matching placebo for dapagliflozin 10 mg
- Balcinrenone/dapagliflozin 40 mg/10 mg (Experimental): Patients will be randomized 1:1:1 to either balcinrenone/dapagliflozin and matching placebo for dapagliflozin or dapagliflozin and matching placebo for balcinrenone/dapagliflozin
  Interventions: Drug: Balcinrenone/dapagliflozin 40 mg/10 mg and matching placebo for dapagliflozin 10 mg
- Dapagliflozin 10 mg (Active Comparator): Patients will be randomized 1:1:1 to either balcinrenone/dapagliflozin and matching placebo for dapagliflozin or dapagliflozin and matching placebo for balcinrenone/dapagliflozin
  Interventions: Drug: Dapagliflozin 10 mg and matching placebo for balcinrenone/dapa gliflozin

INTERVENTIONS:
Drug: Balcinrenone/dapagliflozin 15 mg/10 mg and matching placebo for dapagliflozin 10 mg — 1 capsule of balcinrenone/dapagliflozin 15 mg/10 mg and 1 tablet of matching placebo for dapagliflozin 10 mg once daily, oral use
  Arms: Balcinrenone/dapagliflozin 15 mg/10 mg
Drug: Balcinrenone/dapagliflozin 40 mg/10 mg and matching placebo for dapagliflozin 10 mg — 1 capsule of balcinrenone/dapagliflozin 40 mg/10 mg and 1 tablet of matching placebo for dapagliflozin 10 mg once daily, oral use
  Arms: Balcinrenone/dapagliflozin 40 mg/10 mg
Drug: Dapagliflozin 10 mg and matching placebo for balcinrenone/dapa gliflozin — 1 tablet of dapagliflozin 10 mg and 1 capsule of matching placebo for balcinrenone/dapagliflozin once daily, oral use
  Arms: Dapagliflozin 10 mg

SUMMARY:
The purpose of the study is to evaluate the efficacy, safety and tolerability of balcinrenone/dapagliflozin compared with dapagliflozin alone on patients with chronic kidney disease (CKD) and albuminuria. This study will evaluate the effect of the balcinrenone/dapagliflozin on urinary albumin-to-creatinine ratio (UACR), compared with dapagliflozin in patients with CKD. This is a dose-finding study aiming to identify an optimal dose of balcinrenone/dapagliflozin for a future Phase III study in patients with CKD.

DETAILED DESCRIPTION:
This is a Phase IIb, multicentre, randomised, double-blind, dose-finding, parallel group, double-dummy study aiming to determine the effect on albuminuria, as well as safety and tolerability, of balcinrenone/dapagliflozin compared with dapagliflozin, when given once daily on top of other Standard of Care (SoC) to patients with CKD and albuminuria.

Study population will include participants with CKD (eGFR ≥ 25 to < 60 mL/min/1.73 m2) and UACR > 100 mg/g to ≤ 5000 mg/g. Participants with or without a diagnosis of T2DM and with or without an SGLT2 inhibitor treatment at screening are eligible for the study.

The study will be conducted at approximately 110 sites in approximately 16 countries globally.

At least 300 participants will be randomised in order to have 300 evaluable participants.

Participants will be randomised to one of 3 treatment arms in a 1:1:1 ratio:

* Balcinrenone/dapagliflozin 15 mg/10 mg
* Balcinrenone/dapagliflozin 40 mg/10 mg
* Dapagliflozin 10 mg

For each participant, the total duration of participation will be approximately 23 weeks: an up to 3-week screening period followed by a 12-week treatment period, and an 8-week follow-up period after end of investigational medicinal product (IMP) treatment.

ELIGIBILITY:
Inclusion Criteria: - Age ≥ 18 years old - Diagnosis of CKD and eGFR ≥ 25 to < 60 mL/min/1.73 m2. - UACR > 100 mg/g (10 mg/mmol) to ≤ 5000 mg/g (500 mg/mmol). - Serum potassium ≥ 3.5 mmol/L to ≤ 5.0 mmol/L. - Stable RAAS inhibitors treatment for 4 weeks before screening. Participants who cannot tolerate or are not treated with RAAS inhibitors can also participate in the study. Exclusion criteria: - Uncontrolled arterial hypertension (SBP > 160 mmHg or DBP > 100 mmHg). - Hypotension defined as SBP < 100 mmHg. - Autosomal dominant polycystic kidney disease, lupus nephritis or ANCA-associated vasculitis or other nephropathies that are unstable or progress rapidly. - Cytotoxic or immunomodulatory therapy within 6 months prior to screening, or current, or planned within 6 months following randomization. - History of solid organ or bone marrow transplantation - Recent (90 d prior to screening) or ongoing dialysis, or likely need for dialysis within 3 months following randomization. - Myocardial infarction, acute coronary syndrome, stroke or transient ischaemic attack within the previous 12 weeks. - Type 1 diabetes mellitus (DM) or uncontrolled type 2 DM. - Hepatic disease, including active hepatitis, and/or hepatic impairment (Child-Pugh class B-C; or any of AST or ALT > 3 × ULN; or TBL > 2 × ULN. - Serum HCO3 < 18 mmol/L at screening. - Adrenal insufficiency (eg, Addison's disease, prolonged use of glucocorticoids). - Any use of the following within 4 weeks prior to screening: - MRA (or planned initiation of MRA treatment), potassium sparing diuretic, potassium binders, fludrocortisone. - Strong or moderate CYP3A4 inducers or inhibitors prohibited at least 1 week prior to randomisation and during treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Relative change in UACR from baseline to Week 12 | Baseline (Day 1) until Week 12 (Day 85)
  Evaluating the effect of balcinrenone/dapagliflozin compared with dapagliflozin alone on UACR.

CONTACTS AND LOCATIONS:
Locations (80):
- United States (13):
  - Research Site, Sheffield, Alabama
  - Research Site, Glendale, California
  - Research Site, Waterbury, Connecticut
  - Research Site, Hialeah, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Annapolis, Maryland
  - Research Site, New Bern, North Carolina
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Ogden, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Norfolk, Virginia
- Austria (4):
  - Research Site, Linz
  - Research Site, Sankt Pölten
  - Research Site, Vienna
  - Research Site, Wels
- Brazil (2):
  - Research Site, Porto Alegre
  - Research Site, São Paulo
- Bulgaria (5):
  - Research Site, Burgas
  - Research Site, Dobrich
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
- Canada (4):
  - Research Site, London, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- China (4):
  - Research Site, Changchun
  - Research Site, Changzhou
  - Research Site, Shanghai
  - Research Site, Tianjin
- Italy (5):
  - Research Site, Bari
  - Research Site, Bologna
  - Research Site, Genoa
  - Research Site, Novara
  - Research Site, Pavia
- Japan (11):
  - Research Site, Ageo
  - Research Site, Fujisawa-shi
  - Research Site, Fukuoka
  - Research Site, Koga-shi
  - Research Site, Koshigaya-shi
  - Research Site, Kumamoto
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Okinawa-shi
  - Research Site, Takamatsu
  - Research Site, Zentsuji-shi
- Malaysia (5):
  - Research Site, Ipoh
  - Research Site, Johor Bahru
  - Research Site, Kajang
  - Research Site, Kota Bharu
  - Research Site, Kuala Terengganu
- Poland (6):
  - Research Site, Bialystok
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Leżajsk
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Żywiec
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Palma de Mallorca
  - Research Site, Valencia
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- Turkey (Türkiye) (5):
  - Research Site, Ankara
  - Research Site, Gaziantep
  - Research Site, Kahramanmaraş
  - Research Site, Kayseri
  - Research Site, Kocaeli
- United Kingdom (4):
  - Research Site, Dundee
  - Research Site, London
  - Research Site, Newquay
  - Research Site, Nottingham
- Vietnam (3):
  - Research Site, Haiphong
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Heerspink HJL, Cardona JF, Jolly S, Pergola PE, de Sousa-Amorim E, Eriksson AL, Fredholm M, Gasparyan SB, Guzman NJ, Hartleib-Geschwindner J, Jiang Y, Leonsson-Zachrisson M, Mark PB; MIRO-CKD study investigators. Balcinrenone in combination with dapagliflozin compared with dapagliflozin alone in patients with chronic kidney disease and albuminuria: a randomised, active-controlled double-blind, phase 2b clinical trial. Lancet. 2025 Nov 22;406(10518):2449-2460. doi: 10.1016/S0140-6736(25)02014-8. Epub 2025 Nov 8. PMID 41218621
- [Derived] Mark PB, De Sousa-Amorim E, Eriksson AL, Leonsson-Zachrisson M, Guzman NJ, Miller MT, Jiang Y, Heerspink HJL. Efficacy and safety of balcinrenone and dapagliflozin for CKD: design and baseline characteristics of the MIRO-CKD trial. Nephrol Dial Transplant. 2025 Nov 26;40(12):2280-2288. doi: 10.1093/ndt/gfaf119. PMID 40623005
- [Derived] Bhattacharya CS, Ericsson H, Johansson S, Parkinson J, Boca SM, Yang Y, Heijer M, Housler G, Leonsson-Zachrisson M, Hartleib-Geschwindner J, Pizzato PE. The effect of severe renal impairment on the pharmacokinetics, safety and tolerability of balcinrenone. Br J Clin Pharmacol. 2025 Jul;91(7):1937-1946. doi: 10.1002/bcp.70017. Epub 2025 Feb 17. PMID 39962632